CLINICAL TRIAL: NCT06036914
Title: Ultra High Dose Diuretic Strategy for Management of Acute Decompensated Heart Failure - A Randomized, Double-Blind Pilot Trial
Brief Title: A Study of Ultra High Dose Diuretics to Treat Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yogesh Reddy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-005262
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; With Decompensation
MeSH Terms: conditions — Heart Failure | interventions — Bumetanide; Furosemide; Diuretics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultra-high dose diuretic group (Experimental): Subjects with decompensated heart failure requiring hospitalization will receive IV bumetanide.
  Interventions: Drug: Bumetanide
- Standard dose diuretic group (Active Comparator): Subjects with decompensated heart failure requiring hospitalization will receive IV furosemide.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Bumetanide — Bumetanide will be administered via intravenous (IV) infusion at a dose of 12.5 mg two times a day (BID) for 2 doses total within 24 hours.
  Other Names: Ultra-high dose diuretic
  Arms: Ultra-high dose diuretic group
Drug: Furosemide — Furosemide will be administered via intravenous (IV) infusion at usual doses (twice the home dose of oral daily diuretic in furosemide equivalents) administered as 2 doses total within 24 hours.
  Furosemide equivalents will be considered as follows (40 mg of intravenous furosemide = 1 mg oral bumetanide or 40 mg of torsemide or 80 mg of oral furosemide consistent with prior literature). The lowest dose of furosemide administered during the study will be 40 mg IV two times a day (BID) and the maximum dose will be 100 mg IV BID.
  Other Names: Standard dose diuretic
  Arms: Standard dose diuretic group

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of ultrahigh dose diuretics compared to standard dose diuretics over 24 hours in patients with decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of decompensated heart failure receiving intravenous diuretics
* Ability to provide informed consent

Exclusion Criteria:

* Patients on home inotrope medications
* Patients with Chronic Kidney disease stage V and end stage renal failure on dialysis
* Patients lacking the capacity to consent for themselves
* Known pregnancy or breastfeeding mothers
* Complex congenital heart disease
* Allergy to furosemide or bumetanide
* Respiratory failure requiring non-invasive ventilation (CPAP/BiPAP) or invasive mechanical ventilatory support at the time of randomization
* Hypotension with systolic blood pressure <80 mm Hg at the time of randomization
* Acute coronary syndrome
* Sustained Ventricular tachycardia requiring treatment in the last 48 hours
* Patients weighing ≤ 40 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Reddy, M.B.B.S, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultra-high Dose Diuretic Group: Subjects with decompensated heart failure requiring hospitalization received IV bumetanide.
  Bumetanide: Bumetanide was administered via intravenous (IV) infusion at a dose of 12.5 mg two times a day (BID) for 2 doses total within 24 hours.
- Standard Dose Diuretic Group: Subjects with decompensated heart failure requiring hospitalization received IV furosemide.
  Furosemide: Furosemide was administered via intravenous (IV) infusion at usual doses (twice the home dose of oral daily diuretic in furosemide equivalents) administered as 2 doses total within 24 hours.
  Furosemide equivalents were considered as follows (40 mg of intravenous furosemide = 1 mg oral bumetanide or 40 mg of torsemide or 80 mg of oral furosemide consistent with prior literature). The lowest dose of furosemide administered during the study was 40 mg IV two times a day (BID) and the maximum dose was 100 mg IV BID.
Period: Overall Study
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (12.4) | 70.9 (14.3) | 69 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Urine Output
Description: The total volume of urine produced in milliliters (mL) over 24 hours after initiation of intravenous diuretic.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 9 | 10
mL | 5283 (2976) | 2819 (1060)

2. Secondary Outcome: Change in Body Weight
Description: Change in Body Weight (kg) from Baseline to 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 9 | 10
kg | -2.6 (3.0) | -3.8 (3.3)

3. Secondary Outcome: Change in NT-proBNP
Description: Change in NT-proBNP levels (pg/ml) from Baseline to 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 9 | 10
pg/ml | 2898 (7278) | -1705 (1712)

4. Secondary Outcome: Change in Urine Sodium Excretion
Description: Change in amount of sodium (mmol) excreted in the urine from Baseline to 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: Data for this outcome measure was not collected for any participants. Upon study initiation, this outcome measure was not technically feasible to obtain with existing staffing and was therefore not performed. As a results, no data was collected for this outcome measure.
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Apnea-hypopnea Index
Description: The apnea-hypopnea index (AHI) is the number of apneas and hypopneas per hour of sleep which is an indicator of severity of sleep apnea
  AHI will be measured using a Watch Pat or Nox device at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: Data for this outcome measure was not collected for any participants. Upon study initiation, this outcome measure was not technically feasible to obtain with existing staffing and was therefore not performed. As a result, no data was collected for this outcome measure.
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Iohexol Glomerular Filtration Rate (GFR)
Description: Renal or kidney function was measured by GFR determined by Iohexol clearance. Iohexol GFR will be measured at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: as for outcome 5
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Peripheral Vein Pressure
Description: Peripheral vein pressure (mm Hg) will be recorded from existing IV lines through pressure transducer monitoring at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: Data was not collected for 1 subject in the Ultra-High dose diuretic group as the subject requested that peripheral vein pressure data not be collected on them.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 8 | 10
mmHg | -10.9 (7.5) | -4 (3.1)

8. Secondary Outcome: Change in Cardiac Output
Description: Cardiac output (L/min) is the total volume of blood moved by the heart per minute and will be measured by echocardiography conducted at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: Data was not technically feasible to obtain for 3 subjects in the Ultra-High Dose diuretic group for this outcome measure.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 6 | 10
L/min | -0.53 (0.83) | 0.29 (1.50)

9. Secondary Outcome: Change in Estimated Right Ventricular (RV) Systolic Pressure
Description: Estimated RV systolic pressure (mm Hg) will be measured by echocardiography conducted at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: as for outcome 5
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Right Atrial (RA) Pressure
Description: RA pressure (mm Hg) will be measured by echocardiography conducted at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: as for outcome 5
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Left Atrial (LA) Strain
Description: LA strain will be assessed by echocardiography conducted at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: as for outcome 5
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Left Ventricular (LV) Global Longitudinal Strain
Description: LV global longitudinal strain will be assessed by echocardiography conducted at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: as for outcome 5
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Right Ventricular (RV) Global Longitudinal Strain
Description: RV global longitudinal strain will be assessed by echocardiography conducted at Baseline and 24 hours after initiation of intravenous diuretic.
Time Frame: Baseline, 24 hours
Population: as for outcome 5
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in E/e'
Description: E/e' will be assessed using echocardiography conducted at Baseline and 24 hours after initiation of intravenous diuretic. It is defined as the ratio of peak early diastolic mitral inflow velocity (E) and peak early diastolic mitral annular velocity (e').
Time Frame: Baseline, 24 hours
Population: as for outcome 5
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 90 days.
Description: Adverse events were collected through specific questioning and telephone follow ups.
Arm/Group | Ultra-high Dose Diuretic Group | Standard Dose Diuretic Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT06036914/Prot_SAP_000.pdf